CLINICAL TRIAL: NCT06549699
Title: MUTTON-HF (Medically Used Tailored Traditional Food to Optimize Nutrition) in Heart Failure)
Brief Title: Medically Used Tailored Traditional Food to Optimize Nutrition in Heart Failure
Acronym: MUTTON-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Indian Health Service (IHS) (U.S. Federal Agency); American Heart Association (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08072024
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
Keywords: Indigenous; Navajo; Traditional Foods; Nutrition security; food is medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal delivery program (Active Comparator): Patients will receive 2 meals daily (14 meals weekly) of medically-tailored meals incorporating traditional Navajo foods, followed by a cooking class at the end of the meal program (meals provided for 60 days).
  Interventions: Other: Medically Tailored Meal Program with Traditional Navajo Foods
- Usual Care (Placebo Comparator): Patients will receive usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Medically Tailored Meal Program with Traditional Navajo Foods — Patients will receive medically-tailored meals incorporating local traditional Navajo foods
  Arms: Meal delivery program
Other: Usual Care — Usual care plus healthy recipes provided
  Arms: Usual Care

SUMMARY:
Study subjects with heart failure will receive either pre-prepared, home-delivered DASH/SRD-compliant meals incorporating local Navajo traditional foods or usual care for 60 days (14 meals weekly).

DETAILED DESCRIPTION:
The American Indian and Alaska Native population has experienced significant cardiovascular health disparities compared with other racial and ethnic groups in the U.S. [1] Heart failure, in particular, causes significant morbidity and mortality in Navajo Nation. For many Navajo patients, similar to other American Indian populations, food insecurity is a major driver of health disparities. [2][3] In fact, qualitative data from our heart failure patient advisory committee have found that 89% of patients with heart failure believe nutrition insecurity is a major barrier to optimal health. Dietary factors are believed to be an important cause of hospitalizations in patients with heart failure and cardiovascular outcomes. There is increasing evidence that direct dietary support, such as produce prescription or provision of medically tailored meals may improve cardiovascular outcomes and disease-specific quality of life.[4][5] Furthermore, there has been an increased focus in Indigenous communities to reclaim traditional indigenous foods to improve health. However, more evidence of the benefit of traditional Indigenous foods for cardiovascular health is needed.

The investigators, therefore, in discussion with community members and tribal partners at two Indian Health Service (IHS) sites in Navajo Nation, will implement and evaluate the effectiveness of a medically and Native-sourced culturally tailored meal delivery program to improve outcomes in heart failure in rural Navajo Nation. This study will include two phases, with a phase I pilot feasibility study, followed by phase II-a comparativeness effectiveness randomized control trial to compare the implementation of our medically and culturally tailored meal delivery program compared to usual care. Phase I outcomes will include implementation outcomes such as feasibility and acceptability to inform phase II. The primary outcome for the trial in Phase II will be the proportion of patients who have a hospitalization or ER visit for any cause within 90 days post implementation. Secondary outcomes will include: heart failure hospitalizations specifically, ER visits for volume overload specifically (ER visits for lower extremity edema, dyspnea, with clinical evaluation consistent with volume overload) within 90 days, Kansas City Cardiomyopathy Questionnaire clinical summary score at baseline and at 60 days; prescription adherence rates (% of filled prescriptions out of prescriptions made) for all medication as well as GDMT specifically at 60 days, weight at baseline (and BMI) at 60 days, and the following lab parameters and biomarkers at baseline and at 60 days: albumin, prealbumin, creatinine, NT-proBNP, HbA1c, Total cholesterol, LDL-C, HDL-C, Triglycerides, CRP, and measures of food insecurity. The investigators will also collect measures of Indigenous cultural connectiveness using the validated Cultural Connectedness Scale-California (CCS-CA) at baseline and at 60 days, as well as qualitative analyses of local food suppliers to evaluate how this program strengthens local food systems. The investigators will also evaluate food diaries and perform a survey at 90 days to evaluate for any sustainable change in diet and behavior post intervention. Semi-structured interviews will be performed of stakeholders including a subset of patients, primary care providers and food suppliers to assess implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* ICD I50* diagnosis
* Clinical encounter in last 12 months
* Primary care physician at the two IHS sites
* Hospitalization (any-cause) or ER visit within last 12 months

Exclusion Criteria

* Hospice care
* Living in acute rehabilitation or skilled nursing facility
* Living outside the Gallup Service Unit (outside 50-mile catchment area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization or Emergency Department Visit | 90 days
  Hospitalization or Visit to Emergency Department (All-cause)

SECONDARY OUTCOMES:
Cultural Connectedness Scale-California | 60 days
  The investigators will measure cultural connectedness utilizing a 6-question modified version of the validated Cultural Connectedness Scale-California (CCS-CA) at baseline and at 60 days. This is a validated score, developed by Indigenous scholars to measure cultural connectiveness in Indigenous populations, and has been shown to correlate with physical health and be a social determinant of health. This scale has previously been modified for use in Diné populations specifically by the investigators. The investigators will evaluate total score, as well as subcomponents of identity, traditions, and spirituality.
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 60 days
  This is a validated score for evaluating quality of life and symptom measures in heart failure patients. Score ranges from 0-100, with 0 meaning very poor quality of life/symptoms and health status, 100 meaning excellent quality of life/symptom burden/health status.
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) Quality of Life Subset | 60 days
  Subset of this is a validated score for evaluating quality of life measures in heart failure patients. Score ranges from 0-100, with 0 meaning very poor quality of life/symptoms and health status, 100 meaning excellent quality of life/symptom burden/health status.
Food Security | 60 days
  The investigators will evaluate baseline and 60-day rates of food insecurity utilizing the USDA Adult Food Security: Six Item short Form survey (USDA FSSM 6-Item).[12] At the 60-day evaluation, the investigators will adapt the USDA FSSM 6-Item questionnaire to evaluate food insecurity within the last 2 (rather than 12 months).
Biomarker Data | 60 days
  albumin, prealbumin, creatinine, NT-proBNP, HbA1c, Total cholesterol, LDL-C, HDL-C, Triglycerides, CRP
Weight | 60 days
  Weight (kilograms). Weight and height will be combined to report BMI in kg/m^2
ER visits | 90 days
  All cause
Hospitalizations | 90 days
  All cause
ER visit for Heart Failure | 90 days
  ER visit for volume overload or HF symptoms
Heart Failure hospitalization | 90 days
Diet Quality | 60 Days, 90 days
  The investigators will assess diet quality using the 10-item DSQ [11] with an addition question to assess traditional Diné food intake (During the past month, how often did the participant eat traditional Diné foods (such as blue corn mush, steamed, roasted or dried corn, sumac berries, mutton, local varieties of squash or beans) at baseline and at the end of the intervention.
Financial Stress | 60 Days
  The investigators will measure Financial Stress Scale at baseline and at 60 days using two questions:[16] How worried was the participant over the last 2 months about paying for housing (rent, mortgage, etc.)? How worried was the participant over the last 2 months about paying monthly bills?
  § All questions will be answered on a 4-point scale, where 1 = "not worried at all", 2 = "not too worried", 3 = "moderately worried", and 4 = "very worried"
Intervention characteristics: Partnership | 60 Days
  The investigators will evaluate the following:
  * % of meals that include locally sourced ingredients
  * % of food supply sourced by Diné producers/suppliers/farmers
  * % of meals sourced by Native suppliers/farmers
Implementation Outcomes: Feasibility | 60 Days
  The investigators will evaluate the percentage of meals delivered successfully to the patient (or percentage of meals that were successfully picked up by the patient if picked up from the food pantry or other location).
Implementation Outcomes: Fidelity | 60 Days
  The investigators will assess baseline dietary patterns through 3-day food diaries during week 1 and week 8 after enrollment. The investigators will also survey participants on the % of meals consumed at 60 days. Additionally at 90 days, the investigators will perform a survey to evaluate dietary patterns post intervention and adoption of any of the recipes/behavioral changes.
Implementation Outcomes: Acceptability | 60 Days
  The investigators will evaluate patient satisfaction by evaluating the Net Promoter Score (i.e. how likely is it that the patient would recommend this program to a community member?") post-intervention.
Qualitative Implementation Outcomes: Fidelity, acceptability, feasibility, adoption | 60 Days
  The investigators will perform semi-structured interviews of non-patient stakeholders (i.e. farmers that supplied produce, livestock farmers, food pantry) to assess acceptability and feasibility of providing produce for the meals, as well as the degree to which the program contributed to strengthening the local food system. The investigators will also perform semi-structured interviews of primary care providers and a subset of patients. Semi-structured interviews will be guided by the Consolidated Framework for Implementation Research (CFIR), and the investigators will explore multiple constructs within each CFIR domain that are hypothesized by the study team and based on existing literature to be relevant to acceptability and feasibility of the program.
Physical Activity | 60 Days
  The investigators will evaluate how much physical activity/exercise patients are participating in weekly at baseline, and at 60 days by asking patients to estimate the number of minutes weekly that they are participating in formal exercise or physical activity.
General Health Status | 60 Days
  The investigators will evaluate patients' general health status using a single general health status question (would the patient that in general their health is excellent, very good, good, fair, or poor) at baseline and post-intervention
KCCQ12-PL Physical Limitation Score | 60 Days
  Subsection of KCCQ-12 Score
KCCQ12-SF Symptom Frequency Score | 60 Days
  Subsection of KCCQ12 Score
KCCQ-SL Social Limitation Score | 60 Days
  Subsection of KCCQ-12 Score
Indigenous Nourishment Scale | Baseline, 60 days
  The investigators will evaluate the Indigenous Nourishment Scale (Measure A), which is a scale developed through community-based methods in Indigenous communities to encompass multiple dimensions of nourishment. The investigators will assign score of 0-6 for each response (0 for never-6 for always), for a total score 0-54 (with 0 meaning low levels of nourishment and 54 high levels of nourishment.
Height | 60 days
  Height (cm). Weight and height will be combined to report BMI in kg/m^2.
urine albumin:creatinine | 60 days
  Urine albumin:creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Eberly, MD, MPH, Principal Investigator — Indian Health Service (IHS)
Locations (2):
- United States (2):
  - Gallup Indian Medical Center, Gallup, New Mexico
  - Tohatchi Health Clinic, Tohatchi, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://www.muttonhf.com/